CLINICAL TRIAL: NCT03868020
Title: Pilot Study of 18F Fluciclovine PET CT in Identification of the Primary in Patients With an Unknown Primary Head and Neck Squamous Cell Carcinoma Presenting With Metastatic Cervical Nodal Disease
Brief Title: Fluciclovine F18 PET/CT in Identifying the Origin of Head and Neck Squamous Cell Carcinoma in Patients With Metastatic Cervical Nodal Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-0898; NCI-2019-00597 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0898 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-03-07; First posted 2019-03-08 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Squamous Cell Carcinoma in Cervical Lymph Node
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — fluciclovine F-18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (fluciclovine F18 PET/CT) (Experimental): Patients receive fluciclovine F18 IV and undergo PET/CT scan over 20-30 minutes.
  Interventions: Procedure: Computed Tomography; Radiation: Fluciclovine F18; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Radiation: Fluciclovine F18 — Given IV
  Other Names: (18F)Fluciclovine; (18F)GE-148; 18F-Fluciclovine; [18F]FACBC; Anti-(18f)FABC; Anti-1-Amino-3-[18F]Fluorocyclobutane-1-Carboxylic Acid; Anti-[18F] FACBC; Axumin; Fluciclovine (18F); FLUCICLOVINE F-18; GE-148 (18F); GE-148 F-18
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This early phase I trial studies how well fluciclovine F18 positron emission tomography (PET)/computed tomography (CT) works in identifying the origin of head and neck squamous cell carcinoma in patients with cancer that has spread to the cervical lymph nodes. Fluciclovine F18 during a PET/CT scan may work better in helping doctors learn where the cancer started (called the site of origin) and directing treatment planning compared to standard fludeoxyglucose F-18 (FDG) PET-CT scans.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate positive predictive value with a corresponding 95% confidence interval for fluciclovine F18 (18F fluciclovine) positron emission tomography computed tomography (PET CT) to detect a primary site of disease in patients presenting with cervical metastatic nodal disease but a head and neck primary site not apparent on CT of the neck with contrast (contrast enhanced-computed tomography, CE-CT).

SECONDARY OBJECTIVES:

I. To estimate positive predictive value with a corresponding 95% confidence interval for fludeoxyglucose F-18 (18F FDG) PET CT in the detection of a primary site of disease in patients presenting with cervical metastatic nodal disease but a head and neck primary site not apparent on CT of the neck with contrast.

EXPLORATORY OBJECTIVES:

I. To compare the lesion to background (L/B) ratios for nodal metastatic disease between 18F fluciclovine PET CT and 18F FDG PET CT.

II. To estimate the sensitivity of 18F fluciclovine PET CT and 18F FDG PET CT to detect nodal disease.

III. To evaluate for any trends in findings on 18F fluciclovine PET CT and human papillomavirus (HPV) status.

OUTLINE:

Patients receive fluciclovine F18 intravenously (IV) and undergo PET/CT scan over 20-30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adults with biopsy proven metastatic cervical nodal squamous cell carcinoma
* CT of the neck with contrast that does not confidently identify a primary oropharyngeal site of disease
* Planned standard of care 18F-FDG PET CT examination
* Planned standard of care exam under anesthesia with oropharyngeal surgical biopsy

Exclusion Criteria:

* Pregnant women
* Known allergy to FDG, fluciclovine, or iodine-based contrast agents
* Severe renal dysfunction (glomerular filtrate rate [within 30 days] less than 30)
* Inability to tolerate lying supine, relatively motionless for up to 1 hour

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Proportion of the suspected lesions that are positive by the gold standard of pathology | Up to 2 years
  Positive predicative values will be estimated with a corresponding exact 95% confidence interval.

OTHER OUTCOMES:
Lesion to background (L/B) ratios for nodal metastatic disease | Up to 2 years
  L/B ratios for nodal metastatic disease will be compared between fluciclovine F18 (18F-flucivlovine) positron emission tomography computed tomography (PET CT) and fludeoxyglucose F-18 (18F FDG) PET CT. For lesions that are identified by both 18F FDG PET CT and 18F fluciclovine PET CT, paired t-tests will be used to compare the L/B ratios for primary sites. This analysis will be repeated for nodal metastatic disease sites that are identified by both methods.
Sensitivity and specificity in detecting nodal disease | Up to 2 years
  For nodes that are biopsied, pathology will serve as the gold standard, and the sensitivity and specificity will be estimated separately for 18F FDG PET CT and for 18F fluciclovine PET CT. For nodes that are not, 18F FDG PET CT will serve as the gold standard, and the sensitivity and specificity of 18F-flucivlovine PET CT will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Maria K Gule-Monroe, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org